CLINICAL TRIAL: NCT01885962
Title: Development and Feasibility of an Internet Intervention for Adults With Spinal Cord Injury to Prevent Pressure Ulcers
Acronym: iSHIFTup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Lee M Ritterband, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15409; 10-175 (Other Grant/Funding Number: Virginia Commonwealth Neurotrauma Initiative)
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Spinal Cord Injury; Pressure Ulcers
Keywords: pressure ulcer prevention; spinal cord injury; internet delivered pressure ulcer intervention
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Participants in this group engage in typical rehabilitation and perform usual skin care routine.
- TAU + iSHIFTup (Experimental): Participants in this group engage in typical rehabilitation and use iSHIFTup, Internet Skin Health Intervention for Targeted Ulcer Prevention. Participants are instructed to perform program recommendations to engage in preventive skin care behaviors.
  Interventions: Behavioral: iSHIFTup

INTERVENTIONS:
Behavioral: iSHIFTup — Internet-delivered program to support behaviors to prevent pressure ulcers and promote healthy skin in adults with spinal cord injury.
  Other Names: iSHIFTup, Internet Skin Health Intervention for Targeted Ulcer Prevention
  Arms: TAU + iSHIFTup

SUMMARY:
The investigators propose to test the feasibility of iSHIFTup (Internet Skin Health Intervention For Targeted Ulcer Prevention) for adults with spinal cord injury (SCI) to prevent serious pressure ulcers (PrUs) and promote protective health behaviors. This protocol is Phase 2 of a three phase project. In Phase 1, the investigators developed iSHIFTup. In Phase 2, the investigators will test the intervention by partnering with Woodrow Wilson Rehabilitation Center (WWRC) to conduct a randomized controlled trial (RCT) of 18 participants. In Phase 3, the investigators will focus on optimizing the intervention based on our outcome findings and feedback, sustaining the program at WWRC, and seeking future funding for a larger RCT.

The investigators will conduct an RCT of up to 18 participants (9 participants in treatment as usual (TAU) group, 9 participants in TAU + iSHIFTup intervention group) (18 participants are needed to obtain statistically significant results).

The investigators will meet with potential participants in-person to complete the informed consent process and confirm eligibility. Participants in the TAU+iSHIFTup group will use the program during the study period. Participants randomized to TAU will have usual treatment during the study period and an opportunity to use the program following trial participation. The investigators will collect information from participants at two times during the study, at enrollment and post-intervention at 6-weeks (42 days). The investigators will also collect qualitative information from participants in the TAU+iSHIFTup group, during an optional focus-group setting, to learn users' experiences with the program. The investigators expect participants in the TAU+iSHIFTup group as compared to the TAU group, to display greater awareness of personal risk for pressure ulcers; increased preventive behaviors; and increased skin care self-efficacy and knowledge.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* history of Traumatic Spinal Cord Injury resulting in paraplegia or tetraplegia.
* regular Internet access
* physical ability to use computer
* able to understand, read and speak English
* have identified healthcare provider

Exclusion Criteria:

* SCI of non-traumatic etiology such as:

  * tumor,
  * ischemia,
  * developmental disorders,
  * neurodegenerative diseases,
  * demyelinative diseases,
  * transverse myelitis,
  * vascular malformations.
* Severe pressure ulcer (stage 3 or stage 4).
* Currently pregnant or plan to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Retrospective Diary Data | Baseline and 42 days
  This measure tracks skin care behaviors. It is completed by participants at enrollment and 42 days later. Change in baseline behaviors from baseline to 42 days is measured.
Needs Assessment Checklist (Skin Management Subscale) | Baseline and 42 Days
  Participants complete the NAC-SM after enrollment and again 42 days later. Change in NAC-SM scores from baseline to 42 days is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Ritterband, PhD, Principal Investigator — University of Virginia, Behavioral Health & Technology
Locations (1):
- Woodrow Wilson Rehabilitation Center, Fishersville, Virginia, United States